CLINICAL TRIAL: NCT03456245
Title: A Validation Study of Mobile Technologies for Assessing Visual Acuity and Eye Health Among Older Adults in India
Brief Title: Comparing Low-cost Handheld Autorefractors - a Practical Approach to Measuring Refraction in Low Resource Settings
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Sankara Eye Hospital (Other)
Responsible Party: Principal Investigator, David Bloom, Professor, Harvard School of Public Health (HSPH)
Other Study IDs: 22636
Record Dates: First submitted 2017-07-20; First posted 2018-03-07 (Actual); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Vision device validation: In the single arm of this study, all members of this group were examined using a number of mobile eyesight assessment devices.
  Interventions: Device: Vision device validation

INTERVENTIONS:
Device: Vision device validation — Group members had their vision tested with the following devices/methods: Eyenetra NETRA, PlenOptika Quicksee, Right Manufacturing Retinomax K Plus 3, and standard eyesight tests using eye charts, phoropters, and slit lens lamp imaging.

SUMMARY:
Study compares four portable vision measurement and eye-imaging technologies in terms of accuracy and time and ease of use with older adult (ages 40-100) participants in a developing-country setting (India). Specifically, the five portable devices will be measured against the baseline of the traditional eye-examination techniques, including the use of eye charts and phoropters.

DETAILED DESCRIPTION:
Non-communicable diseases (NCDs) are a large and increasingly costly problem for India. Recent research estimates that NCDs could cost the Indian economy US$6.2 trillion from 2012-2030 if left unaddressed. For some NCDs, new solutions will need to be developed for diagnosis and treatment, while, for others, the necessary interventions exist but are not readily available to all who need them. Visual impairment is one area of health in which limited access to diagnostic and treatment technologies jeopardizes the health and economic well-being of the population. This is particularly true in India, where the population is rapidly aging and, despite the presence of some high-quality medical facilities, there remains a large burden of unaddressed visual impairment.

Loss of visual acuity can negatively impact individual and household income by reducing productivity or hours worked among the visually impaired; it can also affect economic wellbeing via the need for caretakers. There are two key tests that determine visual acuity and measure vision loss:

1. Basic visual acuity (BVA), which is assessed using the naked eye or, when applicable, eyeglasses, and
2. Best-corrected visual acuity (BCVA), which uses refraction to determine eyeglass/contact lens prescription.

In addition, diagnosing vision-hindering eye conditions requires specific medications or surgical procedures. Diagnosis of glaucoma, cataracts, or diabetic retinopathy typically requires a physician to examine a patient's retinas, corneas, and/or pupils at close range using specialized equipment, in conjunction with the visual acuity tests described above.

BCVA tests typically require heavy, cumbersome, and expensive equipment such as phoropters (instruments that measure the refractive state of the eye). Likewise, eye diseases typically require the use of specialized equipment such as slit lamp microscopes, ophthalmoscopes, and tonometers.

However, the recent and anticipated availability of affordable and lightweight portable technologies which can be used both by medical professionals and by trained laypeople has made eye testing easier and faster. This study will validate a number of new handheld devices developed for visual acuity measurement and retinal imaging.

This study explores testing for visual acuity and other impairments like diabetic retinopathy, glaucoma, age-related macular degeneration (AMD), and cataract without the use of traditional stationery and expensive instruments such as phoropters and conventional autorefractors and at a comparatively low cost. If the devices are proven able to accurately evaluate visual acuity and produce high-quality retinal images that can be used to aid diagnosis, it will be a breakthrough in reducing barriers of access to eye care facilities encountered by the majority of the rural population in India and other developing countries.

Also, since these devices are convenient and relatively easy to use, they can be easily used in household/community surveys involving vision measurement; the investigators are proposing to perform data collection for this study in India partially in order to investigate the potential for use of one or more of handheld devices in upcoming waves of the Longitudinal Aging Study in India (Protocol Number 16715), a nationally-representative aging and retirement study that collects data on multiple dimensions of aging, including socioeconomic, cognitive, and health indicators with the aim of informing national policy and practice relating to older adults. Specifically, the study involves an extensive biomarkers module which includes direct measurement of multiple medical and anthropometric indicators, such as blood pressure, grip strength, lung function, height, and weight. The current version of the biomarkers module calls for the use of a traditional eye chart to measure BVA; however, future versions of the study would greatly benefit from the use, if feasible, of portable and inexpensive devices which would allow researchers to collect richer and more accurate data on visual acuity and/or eye conditions and therefore provide a more detailed picture on older adults' eye health, as well as the predictors and correlates of eye health, on a national level.

Through the data gained from this study, the investigators hope to be able to develop useful recommendations for researchers, community health organizations, and health care professionals whose studies and patients would benefit from access to relatively low-cost portable vision measurement and retinal imaging devices. In particular, Indian consumers will have access to all devices pending market approval.

ELIGIBILITY:
Inclusion Criteria:

- Individuals aged 40-100 coming to Sankara Eye Hospital from surrounding urban/rural communities.

Exclusion Criteria:

* Individuals under the age of 40.
* Blind individuals
* Individuals with acute glaucoma, eye trauma/injury, infections such as conjunctivitis
* Individuals physically/cognitively incapable of following basic instructions and sitting/standing still in order to use devices.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged 40-100 coming to Sankara Eye Hospital for standard eyesight evaluation from surrounding urban/rural communities
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E Bloom, PhD, Principal Investigator — Harvard School of Public Health (HSPH)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vision Device Validation: In the single arm of this study, all members of this group were examined using a number of mobile eyesight assessment devices.
  Vision device validation: Group members had their vision tested with the following devices/methods: D-EYE Portable Retinal Imaging System, Eyenetra NETRA, PlenOptika Quicksee, Right Manufacturing Retinomax K Plus 3, and standard eyesight tests using eye charts, phoropters, and slit lens lamp imaging.
Period: Overall Study
Arm/Group | Vision Device Validation
Started | 205
Completed | 190
Not Completed | 15

BASELINE CHARACTERISTICS:
Population: No difference in the population numbers.
Units Other Than Participants: Eyes
Arm/Group | Vision Device Validation
Number analyzed (Participants) | 190
Number analyzed (Eyes) | 374
Age, Continuous [Mean (Full Range); unit: years] | 52.44 [40 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 99
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  India | 190

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Assessment of Participants' Best Visual Acuity (in Diopters)
Description: Measurements of participants' best visual acuity as measured by mobile devices compared to "gold standard" of subjective refraction
Time Frame: 1-2 hours
Population: No difference in the analysis population
Measure: Mean (95% Confidence Interval); unit: Diopters
Arm/Group | Vision Device Validation
Number analyzed (Participants) | 190
Diopters
  Difference btw Subjective refraction and Retinomax | 0.685 [.489 to .881]
  Difference btw Subjective refraction and EyeNetra | -0.416 [-0.675 to -0.157]
  Difference btw Subjective refraction and Quicksee | -0.039 [-0.250 to 0.171]

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Vision Device Validation
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No